CLINICAL TRIAL: NCT04207567
Title: Minute Calisthenics: A Daily, Habit-Based, Bodyweight Resistance-Training Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edward Via Virginia College of Osteopathic Medicine (Other)
Collaborators: Auburn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2019-037
Record Dates: First submitted 2019-12-16; First posted 2019-12-23 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Resistance Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomized (1:1) to an intervention or waitlist control group. The intervention group will perform one set of the bodyweight exercises (i.e., push-ups, angled-rows, bodyweight squats), with training and coaching, unsupervised every weekday for 12 weeks. The waitlist control group will refrain from resistance training for the initial 12.
  After a 12-week follow-up assessment, the intervention group will continue the RT program for an additional 12 weeks, and the waitlist control group will initiate the RT program and continue for 12 weeks. A 24-week follow-up assessment will then be conducted.
Who Masked: Outcomes Assessor
Masking Description: The researchers assessing outcomes as well as the researcher performing statistical analysis will be blinded to participants' group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants in this arm will be instructed to perform one set each of push-ups, angled-rows and bodyweight squats every weekday without supervision for a total of 24 weeks. They will receive the equipment necessary to perform the exercises as well as guidance on proper performance. They will also receive training in the Tiny Habits® Method at baseline and digital coaching for the duration of the study.
  Interventions: Behavioral: Bodyweight exercises (push-ups, angled-rows, bodyweight squats) on weekdays
- Waitlist Control Arm (No Intervention): Participants in the control arm will be instructed to refrain from resistance training for the initial 12 weeks of the study.
  Note that, after the 12-week follow-up assessment (at which the primary outcome of composite reps will be assessed), this group will begin the RT program. They will receive the same equipment, training, and coaching as the intervention group, and they will continue the RT program for 12 weeks, followed by a 24-week assessment.

INTERVENTIONS:
Behavioral: Bodyweight exercises (push-ups, angled-rows, bodyweight squats) on weekdays — Participants will be instructed to perform one set each of push-ups, angled-rows, and bodyweight squats every weekday. They will be given the equipment and training necessary to properly perform the exercises. They will also be trained in the Tiny Habits® Method and receive digital coaching.
  Arms: Intervention Arm

SUMMARY:
As the primary objective, this study will evaluate the effectiveness, in terms of changes in physical strength, of a resistance training (RT) program consisting of brief bodyweight exercises (<5 min/day) performed unsupervised every weekday for 12 weeks. Blood pressure, lipid profile, hemoglobin A1ca, habit strength and satisfaction with the program will also be assessed. Office workers and osteopathic medical students will serve as participants.They will be randomized (1:1) to the intervention group or to a waitlist control group that will refrain from RT for the initial 12 weeks. After the 12-week follow-up assessment, the intervention group will continue the program and the waitlist control group will start the program for 12 weeks, followed by a 24-week follow-up assessment.

DETAILED DESCRIPTION:
Regular resistance training (RT) provides significant health benefits. However, roughly 3 out of 4 US adults do not meet current US Physical Activity Guidelines regarding RT. Studies are needed that assess the effectiveness and feasibility of RT programs that are time-efficient and simple to perform.

This will be a randomized controlled study of a habit-based RT program consisting of one set each of push-ups, angled-rows, and bodyweight squats performed every weekday for 12 weeks. Forty to 60 office workers and osteopathic medical students, who currently do not engage in RT, will be recruited, assessed, and randomized (1:1) to an intervention group, which will perform the exercises as just described, or a waitlist control group, which will refrain from RT for 12 weeks. To promote consistent exercise performance, the intervention group will be trained in the Tiny Habits® Method (a systematic approach to adding new behaviors in one's daily routine) and receive digital coaching for the duration of the study.

After the 12-week follow-up assessment, the intervention group will continue the program for an additional 12 weeks, and the waitlist control group will start the program and continue for 12 weeks, including Tiny Habits training and digital coaching. A 24-week follow-up assessment will then be conducted.

The primary outcome of interest is the change from baseline to 12-weeks in physical strength from, as measured by the maximum number of composite repetitions (i.e., push-ups + angled-rows + bodyweight squats) performed under a standardized protocol. Secondary outcomes of interest include adherence to and satisfaction with the program, and change from baseline to 12- and 24-week follow-up in composite repetitions, habit strength, blood pressure, lipid panel, hemoglobin A1c, body mass index, anthropometry, body composition, and mid-thigh muscle thickness

ELIGIBILITY:
Inclusion Criteria:

* Office worker or osteopathic medical student at the local college/university
* Demonstrate ability to properly perform 1 repetition of each exercise (push-ups, angled-rows, bodyweight squats).
* Indicate having motivation and confidence in ability to perform exercises on weekdays.
* Low adverse event risk while participating, as assessed via the Physical Activity Readiness-Questionnaire (PAR-Q)
* Must be able to identify a suitable location (either at home, school, or office) to set up the suspension system needed to perform the angled-row exercise.

Exclusion Criteria:

* Pregnant
* Participation in structured resistance training for ≥2 days/week, on average, during the past year.
* Implanted medical device (e.g., pacemaker, defibrillator).

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2021-01-04 (Actual)

PRIMARY OUTCOMES:
Physical strength | 12 weeks
  As the primary outcome, the change in physical strength in the intervention group vs. the control group from baseline to 12-week follow-up will be determined by assessing the maximum number of composite repetitions (i.e., push-ups + angled rows + bodyweight squats) that the participant is able to perform under a standardized protocol.

SECONDARY OUTCOMES:
Physical strength | Up to 24 weeks
  The change in physical strength baseline to 24-week follow-up, in the intervention group, and from 12-week follow-up to 24-week follow-up, in the waitlist control group, will be determined by assessing the maximum number of composite repetitions (i.e., push-ups + angled rows + bodyweight squats) that the participant is able to perform under a standardized protocol at those timepoints.
Blood pressure | Baseline, 12-week, and 24-week follow-up
  Measure at baseline, 12-week, and 24-week follow-up following guideline recommendations and using a calibrated automated blood pressure cuff.
Lipid profile | Baseline, 12-week, and 24-week follow-up
  Total cholesterol, (calculated) LDL, HDL, and triglycerides measured at baseline, 12-week, and 24-week follow-up using the CardioChek Plus Analyzer.
Hemoglobin A1c | Baseline, 12-week, and 24-week follow-up
  Measured at baseline, 12-week, and 24-week follow-up using the PTS Diagnostics A1CNow+ System.
Habit strength | 12 weeks
  Each week during the initial 12-weeks of their intervention phase, participants will complete a survey that, among other things, assesses change in habit strength regarding exercise performance (push-ups, angled-rows, bodyweight squats), via the validated Self-Report Behavioral Automaticity Index (SRBAI).
Adherence to protocol | 12 weeks
  Each week during the initial 12-weeks of their intervention phase, participants will complete a survey that, among other things, will assess their (self-reported) adherence to the resistance-training protocol.
Satisfaction with program | 12 weeks
  Each week during the initial 12-weeks of their intervention phase, participants will complete a survey that, among other things, is meant to assess their level of satisfaction with the program.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua C Hollingsworth, PharmD, PhD, Principal Investigator — Edward Via College of Osteopathic Medicine (VCOM-Auburn)
Locations (2):
- United States (2):
  - Auburn University, Auburn, Alabama
  - Edward Via College of Osteopathic Medicine-Auburn Campus, Auburn, Alabama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piercy KL, Troiano RP, Ballard RM, Carlson SA, Fulton JE, Galuska DA, George SM, Olson RD. The Physical Activity Guidelines for Americans. JAMA. 2018 Nov 20;320(19):2020-2028. doi: 10.1001/jama.2018.14854. PMID 30418471
- [Background] National Center for Health Statistics (US). Health, United States, 2017: With Special Feature on Mortality [Internet]. Hyattsville (MD): National Center for Health Statistics (US); 2018. Available from http://www.ncbi.nlm.nih.gov/books/NBK532685/ PMID 30702833
- [Background] Westcott WL. Resistance training is medicine: effects of strength training on health. Curr Sports Med Rep. 2012 Jul-Aug;11(4):209-16. doi: 10.1249/JSR.0b013e31825dabb8. PMID 22777332
- [Derived] Hollingsworth JC, Young KC, Abdullah SF, Wadsworth DD, Abukhader A, Elfenbein B, Holley Z. Protocol for Minute Calisthenics: a randomized controlled study of a daily, habit-based, bodyweight resistance training program. BMC Public Health. 2020 Aug 15;20(1):1242. doi: 10.1186/s12889-020-09355-4. PMID 32799849